CLINICAL TRIAL: NCT05735405
Title: Priming Effects of Aerobic Exercise on Cognitive Training of Patients With Ischemic and Hemorrhagic Stroke
Brief Title: Aerobic Exercise and Cognitive Training in Patients With Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Version 1; 01/09/22
Record Dates: First submitted 2022-11-04; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2022-10

CONDITIONS: Ischemic Stroke; Hemorrhagic Stroke
Keywords: BDNF; Aerobic Exercise; Cognitive Training
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will first perform 30 minutes of pedaling as a moderate intensity aerobic activity. Subsequently it will carry out a daily cognitive training of 60 minutes to improve attentional, working memory and executive functions.
  Interventions: Behavioral: Neuropsychological evaluation; Biological: BDNF evaluation; Behavioral: Pedaling as a moderate intensity aerobic exercise; Other: Cognitive Training; Diagnostic Test: VO2 assessment
- Control Group (Experimental): The control group will first carry out a daily 60-minute cognitive training to improve attentional, working memory and executive functions. It will then perform 30 minutes of pedaling as a moderate intensity aerobic activity.
  Interventions: Behavioral: Neuropsychological evaluation; Biological: BDNF evaluation; Behavioral: Pedaling as a moderate intensity aerobic exercise; Other: Cognitive Training; Diagnostic Test: VO2 assessment

INTERVENTIONS:
Behavioral: Neuropsychological evaluation — Each participant will undergo a complete neuropsychological evaluation, both before and at the end of the clinical trial, with the aim of detecting any changes or improvements.
Biological: BDNF evaluation — During the first and last clinical trial session, each participant will undergo two blood samples, one before and one at the end of the ride, to check levels of Brain Derived Neurotrophic Factor (BDNF).
Behavioral: Pedaling as a moderate intensity aerobic exercise — During each session, each participant will perform 30 minutes of pedaling as a form of moderate intensity physical activity.
Other: Cognitive Training — During each session, each participant will carry out 60 minutes of cognitive training through specific exercises for the attentional, executive and working memory functions.
Diagnostic Test: VO2 assessment — To determine the individual moderate intensity for each patient, a VO2 consumption assessment will be made. The examination will be carried out using an exercise bike and a mask for the calculation of metabolic oxygen consumption.
  The 3 MET threshold to reach in pedaling will be calculated (to define it of moderate intensity), in order to elicit the release of BDNF.

SUMMARY:
The goal of this clinical trial is to test the effects of aerobic exercise and BDNF on patients with ischemic and hemorrhagic stroke during a computerized cognitive training.

The main questions it aims to answer are:

1. Does a moderate intensity aerobic exercise, prior to a cognitive training, allow a better performance?
2. Is it possible to exploit the timing of rehabilitation interventions to obtain greater effects? Participants will be divided in 2 groups. The experimental group will first perform 20 minutes of pedaling as a moderate intensity aerobic exercise. It will then participate in one-hour cognitive training sessions, with the aim of training attentional, working memory and executive functions. The control group will carry out the same interventions but in reverse order.

The researchers will compare the results of the cognitive training in the two groups to verify if the order of the interventions influences the results themselves.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of stroke, both ischemic and haemorrhagic.
* Patients admitted to the Specialist Rehabilitation Unit 1 of the "E. Spalenza - Don Gnocchi "of Rovato.
* Overall score in the MoCA test ³ 26
* In case of a diagnosis of aphasia, a test of verbal comprehension ("Token Test") with score in the norm, P.E. > 1
* Hypertonic and spasticity picture compatible with the performance of motor activity of pedaling expected in the EA session.
* Tolerance of physical exercise
* Incoming electrocardiogram normal and free of anomalies

Exclusion Criteria:

* Overall score in the MoCA test <26
* In case of a diagnosis of aphasia, a test of verbal comprehension ("Token Test") with pathological or borderline score, P.E. £ 1.
* Documented diagnosis of neurodegenerative diseases with impact on performance cognitive.
* Severe acquired brain injury
* Illiteracy
* Status of hypertonus and spasticity not compatible with the performance of motor training
* Excessive fatigue: the patient does not tolerate moderate intensity physical activity and accuses excessive fatigue during the preliminary test
* Electrocardiogram at entrance with anomalies and / or altered
* Ischemic heart disease
* Cardiac disorders that are contraindications for aerobic activity of moderate intensity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-12 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological test scores | Change in the neuropsychological test scores at 1 month
  The experimental hypothesis is to obtain better scores in the experimental group on the neuropsychological tests used. T-tests and delta scores will be used to determine the quantitative change in the score.

SECONDARY OUTCOMES:
Number of errors committed in the cognitive exercises | One month
  For each exercise used in the cognitive training, numerical data will be extrapolated to determine the number of errors committed and the progress achieved. T-tests will be carried out to verify if the experimental group had a better performance during the training than the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Ettore Spalenza- Fondazione Don Gnocchi, Rovato, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Faulkner J, Lambrick D, Kaufmann S, Stoner L. Effects of Upright and Recumbent Cycling on Executive Function and Prefrontal Cortex Oxygenation in Young Healthy Men. J Phys Act Health. 2016 Aug;13(8):882-7. doi: 10.1123/jpah.2015-0454. Epub 2016 May 4. PMID 27144465
- [Background] Abraham WC, Bear MF. Metaplasticity: the plasticity of synaptic plasticity. Trends Neurosci. 1996 Apr;19(4):126-30. doi: 10.1016/s0166-2236(96)80018-x. PMID 8658594
- [Background] Bathina S, Das UN. Brain-derived neurotrophic factor and its clinical implications. Arch Med Sci. 2015 Dec 10;11(6):1164-78. doi: 10.5114/aoms.2015.56342. Epub 2015 Dec 11. PMID 26788077
- [Background] Bediz CS, Oniz A, Guducu C, Ural Demirci E, Ogut H, Gunay E, Cetinkaya C, Ozgoren M. Acute Supramaximal Exercise Increases the Brain Oxygenation in Relation to Cognitive Workload. Front Hum Neurosci. 2016 Apr 20;10:174. doi: 10.3389/fnhum.2016.00174. eCollection 2016. PMID 27148022
- [Background] Borror A. Brain-derived neurotrophic factor mediates cognitive improvements following acute exercise. Med Hypotheses. 2017 Sep;106:1-5. doi: 10.1016/j.mehy.2017.06.024. Epub 2017 Jun 29. PMID 28818262
- [Background] Chang YK, Labban JD, Gapin JI, Etnier JL. The effects of acute exercise on cognitive performance: a meta-analysis. Brain Res. 2012 May 9;1453:87-101. doi: 10.1016/j.brainres.2012.02.068. Epub 2012 Mar 4. PMID 22480735
- [Background] Chmura J, Nazar K, Kaciuba-Uscilko H. Choice reaction time during graded exercise in relation to blood lactate and plasma catecholamine thresholds. Int J Sports Med. 1994 May;15(4):172-6. doi: 10.1055/s-2007-1021042. PMID 8063464
- [Background] Ferris LT, Williams JS, Shen CL. The effect of acute exercise on serum brain-derived neurotrophic factor levels and cognitive function. Med Sci Sports Exerc. 2007 Apr;39(4):728-34. doi: 10.1249/mss.0b013e31802f04c7. PMID 17414812
- [Background] Hennigan A, O'Callaghan RM, Kelly AM. Neurotrophins and their receptors: roles in plasticity, neurodegeneration and neuroprotection. Biochem Soc Trans. 2007 Apr;35(Pt 2):424-7. doi: 10.1042/BST0350424. PMID 17371291
- [Background] Hwang J, Brothers RM, Castelli DM, Glowacki EM, Chen YT, Salinas MM, Kim J, Jung Y, Calvert HG. Acute high-intensity exercise-induced cognitive enhancement and brain-derived neurotrophic factor in young, healthy adults. Neurosci Lett. 2016 Sep 6;630:247-253. doi: 10.1016/j.neulet.2016.07.033. Epub 2016 Jul 20. PMID 27450438
- [Background] Knaepen K, Goekint M, Heyman EM, Meeusen R. Neuroplasticity - exercise-induced response of peripheral brain-derived neurotrophic factor: a systematic review of experimental studies in human subjects. Sports Med. 2010 Sep 1;40(9):765-801. doi: 10.2165/11534530-000000000-00000. PMID 20726622
- [Background] Lambourne K, Tomporowski P. The effect of exercise-induced arousal on cognitive task performance: a meta-regression analysis. Brain Res. 2010 Jun 23;1341:12-24. doi: 10.1016/j.brainres.2010.03.091. Epub 2010 Apr 8. PMID 20381468
- [Background] Nilsson J, Ekblom O, Ekblom M, Lebedev A, Tarassova O, Moberg M, Lovden M. Acute increases in brain-derived neurotrophic factor in plasma following physical exercise relates to subsequent learning in older adults. Sci Rep. 2020 Mar 10;10(1):4395. doi: 10.1038/s41598-020-60124-0. PMID 32157099
- [Background] Rasmussen P, Brassard P, Adser H, Pedersen MV, Leick L, Hart E, Secher NH, Pedersen BK, Pilegaard H. Evidence for a release of brain-derived neurotrophic factor from the brain during exercise. Exp Physiol. 2009 Oct;94(10):1062-9. doi: 10.1113/expphysiol.2009.048512. Epub 2009 Aug 7. PMID 19666694
- [Background] Shobeiri P, Karimi A, Momtazmanesh S, Teixeira AL, Teunissen CE, van Wegen EEH, Hirsch MA, Yekaninejad MS, Rezaei N. Exercise-induced increase in blood-based brain-derived neurotrophic factor (BDNF) in people with multiple sclerosis: A systematic review and meta-analysis of exercise intervention trials. PLoS One. 2022 Mar 3;17(3):e0264557. doi: 10.1371/journal.pone.0264557. eCollection 2022. PMID 35239684
- [Background] Smith PJ, Blumenthal JA, Hoffman BM, Cooper H, Strauman TA, Welsh-Bohmer K, Browndyke JN, Sherwood A. Aerobic exercise and neurocognitive performance: a meta-analytic review of randomized controlled trials. Psychosom Med. 2010 Apr;72(3):239-52. doi: 10.1097/PSY.0b013e3181d14633. Epub 2010 Mar 11. PMID 20223924